CLINICAL TRIAL: NCT02844439
Title: A Phase 2, Multicenter Study of Tesevatinib Monotherapy in Patients With Recurrent Glioblastoma
Brief Title: Study of Tesevatinib Monotherapy in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD019-208
Expanded Access: Available
Record Dates: First submitted 2016-06-24; First posted 2016-07-26 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Glioblastoma (Experimental): The single arm design assessing progression-free survival at 6 months (PFS-6) in the overall population with the ability to detect a rate of 25% is appropriate as a preliminary test of activity in patients with glioblastoma. The sample size of this study is also designed to permit the comparison of results with EGFR amplified and non-amplified tumors, as well as EGFRvIII mutated versus wild-type. The sample size is adequate to characterize the safety profile in patients with glioblastoma.
  Interventions: Drug: Tesevatinib

INTERVENTIONS:
Drug: Tesevatinib
  Other Names: KD019, XL647

SUMMARY:
This is a multicenter, Phase 2 study to assess the activity of tesevatinib in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
This is a multicenter, Phase 2 study to assess the activity of tesevatinib in subjects (n = 40) with recurrent glioblastoma. This study will be conducted at up to 10 sites in the United States.

The availability of paraffin-embedded tumor sample diagnostic of glioblastoma is mandatory for entry into the study. Tumor samples will be evaluated for the EGFRvIII mutation and for EGFR gene amplification. Tissue from recurrent surgery is preferred, but tissue from initial surgery is sufficient for study entry. Baseline MRI is mandatory.

After completion of the screening assessments and confirmation of study eligibility by the Medical Monitor upon review of an inclusion package, tesevatinib will be orally administered to all patients at a dose of 300 mg once daily. A cycle will be considered as 28 days. Patients will be evaluated for efficacy according to the Response Assessment in Neuro-Oncology (RANO) criteria.

Patients who develop ≥ Grade 3 adverse event(s) considered by the investigator to be related to study drug will have study treatment interrupted until the drug-related toxicities have resolved to ≤ Grade 1. Once toxicities have resolved to ≤ Grade 1, the patient may resume study treatment at a reduced dose of 250 mg/day. No more than 1 dose reduction is permitted. Patients who require more than one dose reduction will have study drug discontinued and enter the Follow-up Period.

Patients for whom toxicity persists beyond 21 days despite dose interruption may resume study treatment only with permission from the responsible Medical Monitor.

If study treatment is withheld, the patient should be instructed not to make up the withheld doses.

Study treatment will continue until disease progression, unacceptable toxicity, patient or physician decision to discontinue, or death. Assessments for disease response will occur at Week 4 and Week 8 and then every 8 weeks thereafter using the RANO criteria.

Upon treatment discontinuation, patients will be followed every 8 weeks for survival.

Tumor samples will be used for exploratory biomarker research including, but not limited to, evaluation of EGFRvIII expression by immunohistochemistry or real-time Polymerase Chain Reaction. An appropriate definition and cutoff for EGFRvIII^pos tumors will be established, and outcome in this subpopulation will be evaluated in addition to the overall study population.

To characterize the safety and tolerability profile of tesevatinib, patients will be monitored throughout the study for adverse events (all grades), serious adverse events, and any adverse events requiring drug interruption or discontinuation. Patients will undergo safety evaluations, including physical examinations, Karnofsky Performance Status (KPS), vital sign measurements, hematology, serum chemistry, urinalysis and electrocardiogram.

Magnetic resonance imaging (MRI) will be used to evaluate the tumor at baseline. All MRIs taken on study patients will be submitted to the sponsor for possible retrospective analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide written informed consent and to comply with the study protocol as judged by the investigator
2. Age ≥ 18 years old
3. Kamofsky performance status ≥70%
4. Stable or decreasing dose of corticosteroids within 5 days prior to study 5. enrollment.
5. For women who are not postmenopausal (i.e., < 12 months after last menstruation) or surgically sterile (absence of ovaries and/or uterus) and who are sexually active: agreement to use an adequate method of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly) during the treatment period and for at least 6 months after the last dose of study drug.
6. For male patients who are sexually active and who are partners of premenopausal women: agreement to use a barrier method of contraception during the treatment period and for at least 6 months after the last dose of study drug.
7. Histologically confirmed glioblastoma. A local pathology report constitutes adequate documentation of histology for study inclusion. Patients with an initial diagnosis of a lower-grade glioma are eligible if a subsequent biopsy was determined to be glioblastoma.
8. First recurrence after concurrent or adjuvant chemoradiotherapy. Imaging confirmation of first tumor progression or regrowth as defined by the RANO criteria . A minimum of 12 weeks must have elapsed from the completion of radiotherapy to study entry to minimize the potential for MRI changes related to radiation necrosis that might be misdiagnosed as progression of disease, unless there is a new lesion outside the radiation field or unequivocal evidence of viable tumor on histopathological sampling.
9. Prior treatment with TMZ for low grade glioma or glioblastoma.
10. No more than one prior line of systemic treatment for glioblastoma. Concurrent and adjuvant TMZ-based chemotherapy, including the combination of TMZ with an investigational agent, is considered one line of therapy.
11. Prior therapy with gamma knife or other focal high-dose radiotherapy is allowed, but the patient must have subsequent histologic documentation of recurrence, unless the recurrence is a new lesion outside the irradiated field.
12. Recovery from the toxic effects of prior therapy, with a minimum time of:

    1. ≥ 28 days elapsed from the administration of any prior cytotoxic agents, except ≥ 14 days from vincristine, ≥ 21 days from procarbazine, and ≥ 42 days from nitrosureas
    2. ≥ 28 days elapsed from the administration of any investigational agent
    3. ≥ 14 days elapsed from administration of any non-cytotoxic agent (e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid)
13. Patients who have undergone recent surgery for recurrent or progressive tumor are eligible provided that:

    1. Surgery must have confirmed the recurrence
    2. There must be residual disease
    3. A minimum of 28 days must have elapsed from the day of surgery to first dose of the study drug. For core or needle biopsy, a minimum of 7 days must have elapsed prior to study entry
14. Availability of formalin-fixed paraffin-embedded tumor tissue diagnostic of glioblastoma.

Exclusion Criteria:

1. Concurrent therapeutic intervention (including radiation therapy and NovoTTF).
2. Prior exposure to EGFR inhibitors.
3. Prior exposure to bevacizumab or other VEGF- or VEGF-receptor-targeted agent within 8 weeks of study start.
4. Prior treatment with prolifeprospan 20 with carmustine wafer.
5. Prior intracerebral agent.
6. Evidence of recent hemorrhage on baseline MRI of the brain. However, patients with clinically asymptomatic presence of hemosiderin, resolving hemorrhagic changes related to surgery, or presence of punctuate hemorrhage in the tumor are eligible.
7. Need for urgent palliative intervention for primary disease (e.g., rapidly increasing intracranial pressure, impending herniation, uncontrolled seizures).
8. Hematology:

   ANC < 1.5 x109/L; Plt < 100 x109/L Hgb < 9.0 g/dL within 7 days prior to enrollment. The use of transfusion or other intervention to achieve Hb ≥ 9 g/dL is acceptable.
9. T.Bili. ≥ 1.5 x ULN (except in patients diagnosed with Gilbert's disease).
10. AST(SGOT), ALT(SGPT), or alkaline phosphatase (ALP) ≥ 2.5 x ULN.
11. S. Creat. > 1.5 x ULN.
12. K+ or Mg+ < LLN.
13. In the absence of therapeutic intent to anticoagulate the patient: INR > 1.5 or PT > 1.5 xULN or aPTT > 1.5 xULN Therapeutic anticoagulation.
14. Known contraindication to MRI, such as cardiac pacemaker, shrapnel or ocular foreign body.
15. Used any prescription medication during the prior 2 weeks that the investigator judges is likely to interfere with the study or to pose an additional risk to the patient in participating, specifically inhibitors or inducers of cytochrome P450 (CYP)3A4 (refer to Appendix 5). A stable regimen (≥ 4 weeks) of antidepressants of the selective serotonin re-uptake inhibitor (SSRI) class is allowed (common SSRIs include escitalopram oxalate, citalopram, fluvoxamine, paroxetine, sertraline, and fluoxetine).
16. Taking any drugs associated with torsades de pointes or known to moderately or severely prolong the QTc(F) interval
17. History of torsades de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 50 bpm), heart block (excluding first degree block, being PR interval only), or congenital long QT syndrome. Patients with a history of atrial arrhythmias should be discussed with the Medical Monitor.
18. Uncontrolled diabetes, as evidenced by fasting serum glucose level >200 mg/dL
19. New York Heart Association (NYHA) Grade II or greater congestive cardiac failure.
20. Has marked prolongation of QTc(F) interval at screening or baseline (QTc[F] interval > 470 msec) using the Fridericia method of correction for heart rate.
21. History of myocardial infarction (within 12 months) or unstable angina (within 6 months) prior to study enrolment.
22. History of stroke or transient ischemic attacks within 6 months prior to study enrolment.
23. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study enrolment.
24. Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
25. History of intracranial abscess within 6 months prior to study enrolment.
26. History of another malignancy in the previous 3 years, with a disease-free interval of < 3 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible.
27. Evidence of any active infection requiring hospitalization or IV antibiotics within 2 weeks prior to study enrolment.
28. Known hypersensitivity to any excipients of tesevatinib.
29. Inability to swallow or absorb orally-administered medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Center for Neurosciences, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - UT MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects at least 18 years of age with recurrent glioblastoma and no concurrent therapeutic intervention including prior exposure to EGFR inhibitors, VEGF, carmustine wafer, or intracerebral agent
Pre-assignment Details: A total of 40 subjects with recurrent glioblastoma were enrolled. Tumor samples were evaluated for the presence or absence of EGFR gene-amplification, designated Sub-population A, and/or the EGFR variant III mutation (EGFRvIII^pos), designated Sub-population B, or neither EGFR gene-amplification nor EGFRvIII^pos variant mutation.
  Note: EGFR = epidermal growth factor receptor; EGFR vIII^pos = EGFR variant 3 mutation; VEGF = vascular endothelial growth factor
Groups:
- Total: Subjects with recurrent glioblastoma who had or did not have EGFR gene-amplified and/or EGFRvIII^pos glioblastoma
Period: Overall Study
Arm/Group | Total
Started | 40 (All Subjects with Glioblastoma: 24 subjects with EGFR-gene amplified + 16 subjects without EGFR gene-amplified nor EGFRvIII^pos)
Subpopulation A (EGFR Gene Amplified Glioblastoma) | 24
Subpopulation B (EGFRvIII^Pos Glioblastoma) | 11
Completed | 0
Not Completed | 40
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Termination by Sponsor | 4
Not completed — Death | 28
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant Sub-population A: With EGFR gene-amplified only Sub-population B: With EGFR gene-amplified + EGFRvIII^pos variant (Subset of Sub-population A) Note: EGFR = epidermal growth factor receptor
Groups:
- Total: All Subjects: Subjects with recurrent glioblastoma who had or did not have EGFR gene-amplified glioblastoma and/or EGFRvIII^pos variant
Arm/Group | Total: All Subjects
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Years
    All Subjects | 55.9 (9.88)
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A | 55.9 (8.37)
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B | 56.8 (8.49)
Age, Customized [Median (Full Range); unit: Years] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Years
    All Subjects | 58.0 [34 to 73]
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A | 57.5 [37 to 73]
    Sub-population B | 58.0 [37 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Participants
    All Subjects: Female | 12
    All Subjects: Male | 28
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: Female | 6
    Sub-population A: Male | 18
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: Female | 3
    Sub-population B: Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Participants
    All Subjects: Hispanic or Latino | 2
    All Subjects: Not Hispanic or Latino | 37
    All Subjects: Unknown or Not Reported | 1
    Sub-population A (EGFRvIII^pos glioblastoma): number analyzed (Participants) | 24
    Sub-population A (EGFRvIII^pos glioblastoma): Hispanic or Latino | 0
    Sub-population A (EGFRvIII^pos glioblastoma): Not Hispanic or Latino | 23
    Sub-population A (EGFRvIII^pos glioblastoma): Unknown or Not Reported | 1
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: Hispanic or Latino | 0
    Sub-population B: Not Hispanic or Latino | 11
    Sub-population B: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Participants
    All Subjects: American Indian or Alaska Native | 0
    All Subjects: Asian | 4
    All Subjects: Native Hawaiian or Other Pacific Islander | 0
    All Subjects: Black or African American | 1
    All Subjects: White | 34
    All Subjects: More than one race | 0
    All Subjects: Unknown or Not Reported | 1
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: American Indian or Alaska Native | 0
    Sub-population A: Asian | 3
    Sub-population A: Native Hawaiian or Other Pacific Islander | 0
    Sub-population A: Black or African American | 0
    Sub-population A: White | 21
    Sub-population A: More than one race | 0
    Sub-population A: Unknown or Not Reported | 0
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: American Indian or Alaska Native | 0
    Sub-population B: Asian | 2
    Sub-population B: Native Hawaiian or Other Pacific Islander | 0
    Sub-population B: Black or African American | 0
    Sub-population B: White | 9
    Sub-population B: More than one race | 0
    Sub-population B: Unknown or Not Reported | 0
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — Population: Karnofsky Performance Score: 50 = requires considerable assistance and frequent medical care; 60 - requires occasional assistance, but is able to care for most of his personal needs; 70 = cares for self but is unable to carry on normal activity or to do active work; 80 = normal activity with effort and some signs or symptoms of disease; 90 - able to carry on normal activity and minor signs of symptoms of disease; 100 = normal no complaints with no evidence of disease
  Participants
    All Subjects: 50 (Score) | 0
    All Subjects: 60 (Score) | 0
    All Subjects: 70 (Score) | 6
    All Subjects: 80 (Score) | 15
    All Subjects: 90 (Score) | 19
    All Subjects: 100 (Score) | 0
    Sub-population A (EGFRvIII^pos glioblastoma): number analyzed (Participants) | 24
    Sub-population A (EGFRvIII^pos glioblastoma): 50 (Score) | 0
    Sub-population A (EGFRvIII^pos glioblastoma): 60 (Score) | 0
    Sub-population A (EGFRvIII^pos glioblastoma): 70 (Score) | 3
    Sub-population A (EGFRvIII^pos glioblastoma): 80 (Score) | 10
    Sub-population A (EGFRvIII^pos glioblastoma): 90 (Score) | 11
    Sub-population A (EGFRvIII^pos glioblastoma): 100 (Score) | 0
    Sub-population: number analyzed (Participants) | 11
    Sub-population: 50 (Score) | 0
    Sub-population: 60 (Score) | 0
    Sub-population: 70 (Score) | 1
    Sub-population: 80 (Score) | 4
    Sub-population: 90 (Score) | 6
    Sub-population: 100 (Score) | 0
Prior Low Grade Astrocytoma Diagnosis [Count of Participants; unit: Participants] — Population: Low-grade astrocytoma (diffuse astrocytoma): usually an infiltrating tumor that grows relatively slowly and usually does not have well-defined borders
  Participants
    All Subjects: Yes | 2
    All Subjects: No | 38
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: Yes | 0
    Sub-population A: No | 24
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: Yes | 0
    Sub-population B: No | 11
Months Since First Diagnosis of Glioblastoma: Mean [Mean (Standard Deviation); unit: Months] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Months
    All Subjects | 12.59 (8.658)
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A | 13.50 (10.032)
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B | 13.15 (9.010)
Months Since First Diagnosis of Glioblastoma: Median [Median (Full Range); unit: Months] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Months
    All Subjects | 9.95 [1.3 to 47.2]
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A | 8.50 [5.9 to 47.2]
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B | 8.50 [5.9 to 31.7]
Months Since Recurrent Diagnosis of Glioblastoma: Mean [Mean (Standard Deviation); unit: Months] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Months
    All Subjects | 1.34 (2.123)
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A | 1.58 (2.707)
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B | 1.14 (0.916)
Months Since Recurrent Diagnosis of Glioblastoma: Median [Median (Full Range); unit: Months] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Months
    All Subjects | 0.90 [0.2 to 13.8]
    Sub-population A (EGFRvIII^pos glioblastoma): number analyzed (Participants) | 24
    Sub-population A (EGFRvIII^pos glioblastoma) | 0.80 [0.2 to 13.8]
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B | 0.80 [0.2 to 2.7]
Number of Prior Systemic Therapy Regimens [Count of Participants; unit: Participants] — Population: Data were not available for all subjects
  Participants
    All Subjects: 1 Regimen | 21
    All Subjects: 2 Regimens | 16
    All Subjects: > 2 Regimens | 2
    All Subjects: No Prior Systemic Therapy | 1
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: 1 Regimen | 13
    Sub-population A: 2 Regimens | 11
    Sub-population A: > 2 Regimens | 0
    Sub-population A: No Prior Systemic Therapy | 0
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: 1 Regimen | 5
    Sub-population B: 2 Regimens | 6
    Sub-population B: > 2 Regimens | 0
    Sub-population B: No Prior Systemic Therapy | 0
Prior Surgery [Count of Participants; unit: Participants] — Population: All Subjects: With or without EGFR gene-amplified and/or EGFRvIII^pos variant. Sub-population A: EGFR gene-amplified. Sub-population B: EGFRvIII^pos variant (Subset of Sub-population A).
  Participants
    All Subjects: Yes | 39
    All Subjects: No | 0
    All Subjects: Unknown | 1
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: Yes | 24
    Sub-population A: No | 0
    Sub-population A: Unknown | 0
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: Yes | 11
    Sub-population B: No | 0
    Sub-population B: Unknown | 0
Prior Radiotherapy--Site Irradiated [Count of Participants; unit: Participants] — Population: Analysis is for Sub-populations A and B, and for total which includes subjects in both Sub-populations A and B, and neither sub-population.
  Participants
    All Subjects: Brain | 29
    All Subjects: Other | 11
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: Brain | 17
    Sub-population A: Other | 7
    Sub-population: number analyzed (Participants) | 11
    Sub-population: Brain | 7
    Sub-population: Other | 4
Best Overall Response [Count of Participants; unit: Participants] — Best overall response to previous therapy Population: Response Criteria in Solid Tumors (RECIST): CR = complete response; PR = partial response; SD = stable disease; PD = progressive disease;
  Participants
    All Subjects: CR | 0
    All Subjects: PR | 0
    All Subjects: SD | 21
    All Subjects: PD | 9
    All Subjects: Unknown | 10
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: CR | 0
    Sub-population A: PR | 0
    Sub-population A: SD | 12
    Sub-population A: PD | 6
    Sub-population A: Unknown | 6
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: CR | 0
    Sub-population B: PR | 0
    Sub-population B: SD | 5
    Sub-population B: PD | 1
    Sub-population B: Unknown | 5
Reason Therapy Ended [Count of Participants; unit: Participants] — Population: Analysis is for Sub-populations A and B, and for total which includes subjects in both Sub-populations A and B, and neither sub-population.
  Participants
    All Subjects: number analyzed (Participants) | 39
    All Subjects: Treatment Completed | 11
    All Subjects: Progressive Disease | 24
    All Subjects: Study Drug Toxicity | 1
    All Subjects: Other | 3
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: Treatment Completed | 8
    Sub-population A: Progressive Disease | 13
    Sub-population A: Study Drug Toxicity | 1
    Sub-population A: Other | 2
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: Treatment Completed | 5
    Sub-population B: Progressive Disease | 4
    Sub-population B: Study Drug Toxicity | 1
    Sub-population B: Other | 1
Corticosteroid Used at Baseline [Count of Participants; unit: Participants] — Population: Data only available for 4 subjects
  Participants
    All Subjects: None | 3
    All Subjects: Dose increased | 0
    All Subjects: Dose decreased | 0
    All Subjects: Dose stable | 1
    All Subjects: Unknown | 36
    Sub-population A: number analyzed (Participants) | 24
    Sub-population A: None | 2
    Sub-population A: Dose increased | 0
    Sub-population A: Dose decreased | 0
    Sub-population A: Dose stable | 1
    Sub-population A: Unknown | 21
    Sub-population B: number analyzed (Participants) | 11
    Sub-population B: None | 0
    Sub-population B: Dose increased | 0
    Sub-population B: Dose decreased | 0
    Sub-population B: Dose stable | 1
    Sub-population B: Unknown | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Median Progression-free Survival (PFS) Rate at 6 Months (PFS-6)
Description: Proportion (%) of subjects who did not have progressive disease after treatment with tesevatinib at 6 months (PFS-6) after baseline
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage (%) of subjects
Groups:
- Total: Subjects with recurrent glioblastoma who had or did not have EGFR gene-amplified and/or EGFRvIII^pos variant
- Sub-population A: Subjects with EGFR gene-amplified glioblastoma
- Sub-population B: Subjects with EGFR gene-amplified and EGFRvIII^pos variant glioblastoma (Subset of Sub-population A)
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Percentage (%) of subjects | 22.5 [10.8 to 38.5] | 25.0 [9.8 to 46.7] | 18.2 [2.3 to 51.8]

2. Secondary Outcome: Efficacy: Median PFS
Description: Median duration (months) of subjects who were progression-free of disease from baseline
Time Frame: Until disease progression, unacceptable toxicity, subject or clinician decision to discontinue, death, or up to 3 years, whichever occurred first
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Sub-population B: Subjects with EGFR gene-amplified and EGFRvIII^pos glioblastoma (Subset of Sub-population A)
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Months | 2.3 [1.08 to 2.96] | 1.7 [0.95 to 2.96] | 1.0 [0.92 to 4.93]

3. Secondary Outcome: Efficacy: Median Overall Survival Rate at 9 Months (OS-9)
Description: Median proportion (%) of subjects who survived 9 months after baseline
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: Percentage (%) of subjects
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Percentage (%) of subjects | 42.5 [27.0 to 59.1] | 37.5 [18.8 to 59.4] | 27.3 [6.0 to 61.0]

4. Secondary Outcome: Efficacy: Median OS
Description: Median duration (months) subjects survived from baseline until death
Time Frame: Until unacceptable toxicity, subject or investigator decision to discontinue, death, or up to 3 years, whichever occurred first
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Months | 8.4 [7.36 to 12.29] | 7.8 [6.64 to 15.67] | 7.6 [4.93 to 16.62]

5. Secondary Outcome: Efficacy: Best Overall Response
Description: Best overall response that subjects had to treatment with tesevatinib: complete response (CR), partial response (PR), stable disease (SD), or non-response/progressive disease (PD)
Time Frame: Until disease progression, unacceptable toxicity, subject or investigator decision to discontinue, death, or up to 3 years, whichever occurred first
Population: Note: NA = data not available; NE = not evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Participants
  CR | 0 | 0 | 0
  PR | 1 | 1 | 1
  SD | 22 | 10 | 2
  PD | 13 | 10 | 6
  NE | 1 | 1 | 1
  NA | 3 | 2 | 1

6. Secondary Outcome: Efficacy: Objective Response Rate (ORR)
Description: Proportion (%) of subjects who had either a complete response (CR) or a partial response (PR) to treatment with tesevatinib
Time Frame: Until disease progression, unacceptable toxicity, subject or investigator decision to discontinue, death, or 3 years, whichever occurred first
Measure: Number (95% Confidence Interval); unit: Percentage (%) of participants
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Percentage (%) of participants | 2.5 [0 to 13.0] | 4.2 [0 to 21] | 9.1 [0 to 41]

7. Secondary Outcome: Exposure to Tesevatinib: Overall Mean
Description: Mean total amount of tesevatinib (mg) subjects received during the study
Time Frame: Until disease progression, unacceptable toxicity, subject or investigator decision, death, or up to 3 years, whichever occurred first
Measure: Mean (Standard Deviation); unit: mg (tesevatinib)
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
mg (tesevatinib) | 26670.0 (44533.38) | 21752.1 (34748.96) | 11481.8 (7024.22)

8. Secondary Outcome: Exposure to Tesevatinib: Overall Median
Description: Median amount of tesevatinib (mg) subjects received during the study
Time Frame: as for outcome 7
Measure: Median (Full Range); unit: mg (tesevatinib)
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
mg (tesevatinib) | 11850.0 [3900 to 210850] | 10350.0 [4500 to 179150] | 8700.0 [4500 to 25500]

9. Secondary Outcome: Exposure to Tesevatinib: Mean Number of Cycles
Description: Mean number of 28-day cycles of treatment with tesevatinib subjects received during the study
Time Frame: as for outcome 7
Measure: Mean (Standard Deviation); unit: Number of cycles
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Number of cycles | 3.8 (6.72) | 3.3 (6.26) | 1.8 (1.54)

10. Secondary Outcome: Exposure to Tesevatinib: Median Number of Cycles
Description: Median number of 28-day cycles of treatment with tesevatinib subjects received during the study
Time Frame: as for outcome 7
Measure: Median (Full Range); unit: Number of cycles
Arm/Group | Total | Sub-population A | Sub-population B
Number analyzed (Participants) | 40 | 24 | 11
Number of cycles | 2.0 [1 to 32] | 1.5 [1 to 32] | 1.0 [1 to 6]

ADVERSE EVENTS:
Time Frame: Subjects were followed for treatment-emergent adverse events and other safety assessments from screening through 30-day follow-up.
Groups:
- Total: Subjects with recurrent glioblastoma who had or did not have EGFR gene-amplified and/or EGFRvIII^pos variant glioblastoma. Includes 24 subjects who had EGFR gene-amplified (Sub-population A, 11 subjects who had EGFRvIII^pos and EGFR gene-amplified (Sub-population B which is a subset of Sub-population A) and 16 subjects who were in neither sub-population
- Sub-population B: Subjects with EGFRvIII^pos variant glioblastoma (Subset of Sub-population A)
Arm/Group | Total | Sub-population A | Sub-population B
All-Cause Mortality (participants affected / at risk) | 28/40 | 19/24 | 9/11
Serious Adverse Events (participants affected / at risk) | 12/40 | 7/24 | 2/11
Other Adverse Events (participants affected / at risk) | 40/40 | 24/24 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=40) | Sub-population A (N=24) | Sub-population B (N=11)
Hemiparesis (Nervous system disorders) | 2 | 2 | 0
Brain edema (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 1 | 1
Facial paralysis (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 1
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 1
Wound dehiscene (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=40) | Sub-population A (N=24) | Sub-population B (N=11)
Diarrhea (Gastrointestinal disorders) | 31 | 20 | 11
Nausea (Gastrointestinal disorders) | 6 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1
GERD (Gastrointestinal disorders) | 3 | 2 | 1
Anal incontinence (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 2 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 17 | 11 | 5
Rash (Skin and subcutaneous tissue disorders) | 13 | 8 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Aphasia (Nervous system disorders) | 7 | 5 | 1
Hemiparesis (Nervous system disorders) | 7 | 4 | 1
Headache (Nervous system disorders) | 5 | 4 | 2
Dizziness (Nervous system disorders) | 5 | 2 | 0
Seizure (Nervous system disorders) | 5 | 2 | 1
Paresthia (Nervous system disorders) | 3 | 3 | 1
Brain edema (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0 | 0
Facial paresis (Nervous system disorders) | 2 | 2 | 1
Memory impairment (Nervous system disorders) | 2 | 2 | 0
Fatigue (General disorders) | 17 | 9 | 5
Gait disturbance (General disorders) | 6 | 4 | 3
Asthenia (General disorders) | 4 | 2 | 0
Peripheral edema (General disorders) | 3 | 2 | 1
Pain (General disorders) | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 8 | 6 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 5 | 0
QT interval prolongation (Investigations) | 7 | 2 | 0
Weight decreased (Investigations) | 5 | 2 | 1
Hemoglobin decreased (Investigations) | 2 | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 2 | 1
Platelet count decreased (Investigations) | 2 | 2 | 0
Weight increased (Investigations) | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 4 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 1
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Vision blurred (Eye disorders) | 3 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 3 | 2
Hypertension (Vascular disorders) | 3 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 1
Cushingoid (Endocrine disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT02844439/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT02844439/SAP_001.pdf